CLINICAL TRIAL: NCT05337878
Title: A Randomized Double-blind, Placebo-controlled, Non-confirmatory Study to Assess Safety, Tolerability, PK, and PD of Single Ascending and Multiple Doses of ISIS 681257 in Healthy Japanese Participants
Brief Title: A Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Pelacarsen (ISIS 681257) in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: AKCEA-CS1
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Healthy Participants
MeSH Terms: interventions — pelacarsen; AKCEA-APO(a)-LRx

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- SAD: Placebo (Placebo Comparator): Single dose of Pelacarsen-matching placebo administered by SC injection on Day 1 of single-dose treatment period.
  Interventions: Drug: Placebo
- SAD: Pelacarsen 20 milligrams (mg) (Experimental): Single dose of Pelacarsen, 20 mg, administered by SC injection on Day 1 of single-dose treatment period.
  Interventions: Drug: Pelacarsen
- SAD: Pelacarsen 40 mg (Experimental): Single dose of Pelacarsen, 40 mg, administered by SC injection on Day 1 of single-dose treatment period.
  Interventions: Drug: Pelacarsen
- SAD: Pelacarsen 80 mg (Experimental): Single dose of Pelacarsen, 80 mg, administered by SC injection on Day 1 of single-dose treatment period.
  Interventions: Drug: Pelacarsen
- MD: Placebo (Placebo Comparator): Multiple doses of Pelacarsen-matching placebo administered by SC injection every 4 weeks, on Days 1, 29, 57 and 85 of multiple-dose treatment period.
  Interventions: Drug: Placebo
- MD: Pelacarsen 80 mg (Experimental): Multiple doses of Pelacarsen, 80 mg, administered by SC injection every 4 weeks, on Days 1, 29, 57 and 85 of multiple-dose treatment period.
  Interventions: Drug: Pelacarsen

INTERVENTIONS:
Drug: Placebo — Pelacarsen-matching placebo administered by SC injection.
  Arms: MD: Placebo; SAD: Placebo
Drug: Pelacarsen — Pelacarsen administered by SC injection.
  Other Names: AKCEA-APO(a)-LRx; TQJ230; ISIS 681257
  Arms: MD: Pelacarsen 80 mg; SAD: Pelacarsen 20 milligrams (mg); SAD: Pelacarsen 40 mg; SAD: Pelacarsen 80 mg

SUMMARY:
The purpose of the study is to assess the safety, tolerability, and pharmacokinetics (PK) of single and multiple subcutaneous (SC) doses of Pelacarsen (ISIS 681257) in healthy Japanese participants.

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, participant and investigator-blinded, single ascending and multiple-dose study of Pelacrsen (ISIS 681257) in up to 29 healthy Japanese male and female participants. The study was conducted in two parts:1) Single ascending dose (SAD) including up to a 28-day screening period, a baseline period, dose with study drug on Day 1, a 2-day (48 hours) post-dose in-patient observation period, followed by an out-patient observation period up to Day 90; 2) Multiple doses (MD) including up to a 28-day screening period, a baseline period, dose with study drug up to Day 85, a 2-day (48 hours) post-dose in-patient observation period, followed by an out-patient observation period up to Day 204.

In the SAD period, participants were randomized to receive single dose of Pelacarsen or placebo.

Upon completion of the SAD period participants were randomized to receive multiple doses of Pelacarsen.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent (signed and dated) and any authorizations required by local law and was able to comply with all study requirements.
2. Male and female of first-, second- or third-generation Japanese participants.
3. Japanese healthy or obese male and female participants 18 to 65 years of age inclusive, and in good health as determined by past medical history, physical examination, vital signs, ECG and laboratory tests at screening.
4. Participants weighed at least 45 kilograms (kg), healthy or obese with body mass index (BMI) ≤ 35.0 kilograms per meter square (kg/m^2).
5. Participants had to have lipoprotein(a) (Lp[a]) ≥ 15 nanomole per liter (nmol/L) (8 milligram per deciliter [mg/dL]) at screening.

Exclusion Criteria:

1. Clinically significant abnormalities in medical history including acute coronary syndrome, major surgery within 3 months of screening, planned surgery that would have occurred during the study or physical examination or other screening results such as ECGs findings at screening.

Screening laboratory results as follows or any other clinically significant abnormalities in screening laboratory values that would have rendered a participant unsuitable for inclusion. If abnormal, the laboratory tests may have been repeated after consultation with the Sponsor Medical Monitor.

* Estimated glomerular filtration rate (eGFR) ˂ 60 milliliter per minute per 1.73 meter per square (mL/min/1.73m^2) (as determined by the Chronic Kidney Disease-Epidemiological Collaboration [CKD-EPI] Equation).
* Urine protein-to-creatinine ratio (UPCR) ≥ 200 milligram per gram (mg/g) or urine albumin-to-creatinine ratio (UACR) ≥ 30 mg/g.
* Alanine aminotransferase (ALT; serum glutamic pyruvic transaminase), aspartate aminotransferase (AST; serum glutamic oxaloacetic transaminase), bilirubin, alkaline phosphatase, serum creatinine, blood urea nitrogen > 1.5 × upper limit of normal (ULN) at screening excluded a participant from participation in the study.
* Fasting blood glucose > ULN. If elevated, hemoglobin A1c was checked and if < 6%, the participant could have been enrolled.
* Platelet count < 140,000 per microliter (/μL). 3. Active infection requiring systemic antiviral or antimicrobial therapy that would not have been completed prior to Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
SAD: Percentage of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Evaluation Parameters | Up to Day 90
SAD: Percentage of Participants With Adverse Events | Up to Day 90
SAD: Percentage of Participants With Serious Adverse Events | Up to Day 90
MAD: Percentage of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Evaluation Parameters | Up to Day 204
MAD: Percentage of Participants With Adverse Events | Up to Day 204
MAD: Percentage of Participants With Serious Adverse Events | Up to Day 204

SECONDARY OUTCOMES:
Maximum Observed Drug Concentration (Cmax) in Plasma After Single Ascending Dose of Pelacarsen | Day 1: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 up to 168 hours post-dose
Area Under Curve (AUC) From Time Zero to the Last Quantifiable Concentration (AUClast) in Plasma After Single Ascending Dose of Pelacarsen | Day 1: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 up to 168 hours post-dose
Maximum Observed Drug Concentration (Cmax) in Plasma After Multiple Doses of Pelacarsen | Days 1 and 85: Pre-dose; 1, 2, 4, 8, 24 up to 168 hours post-dose
Area Under Curve (AUC) From Time Zero to the Last Quantifiable Concentration (AUClast) in Plasma After Multiple Doses of Pelacarsen | Days 1 and 85: Pre-dose; 1, 2, 4, 8, 24 up to 168 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milosavljevic MN, Stefanovic SM, Pejcic AV. Potential Novel RNA-Targeting Agents for Effective Lipoprotein(a) Lowering: A Systematic Assessment of the Evidence From Completed and Ongoing Developmental Clinical Trials. J Cardiovasc Pharmacol. 2023 Jul 1;82(1):1-12. doi: 10.1097/FJC.0000000000001429. PMID 37070852